CLINICAL TRIAL: NCT06801080
Title: Well Baby, Well Family Study
Acronym: WBWF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Naval Health Research Center (U.S. Federal Agency)
Collaborators: Abt Global (Unknown)
Responsible Party: Principal Investigator, Jessica Redding, Compliance administrator, Deployment Health Department, Naval Health Research Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NHRC.2019.0021
Record Dates: First submitted 2025-01-21; First posted 2025-01-30 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Social Determinants of Health
Keywords: HealthySteps; New parent support; military children; social determinants of health
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This was a quasi-experimental study of military parents with a newborn infant seeking care at DoD HS pilot program implementation pediatric clinics as well as pediatric clinics at military treatment facilities implementing treatment as usual. The target population included parents with an infant aged 0-4 months scheduling well-baby care at one of 7 pilot and 11 comparison clinics. Participation in both the HS pilot services and the WBWF study was voluntary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HealthySteps Pilot (Experimental): The intervention arm included 3 tiers of targeted care following the HS model (https://www.zerotothree.org/our-work/healthysteps/). At tier 1, the standard Bright Futures screenings used in DoD pediatrics for children age 0 to 3 years were augmented to assess child social emotional development and family needs. For tiers 2 and 3, pediatricians/medical staff could refer eligible families with children aged 0 to 3 years to a HS Specialist either to address a specific issue requiring time-limited services (tier 2) or for comprehensive services (tier 3) to receive support at all well-child visits. Further, to meet the requirements of NDAA FY19, section 578, the HS Specialists were instructed to offer tier 3 services to all families of infants aged 0-4 months; this population was the WBWF intervention population eligible for the intervention arm of this study.
  Interventions: Other: HealthySteps (https://www.zerotothree.org/our-work/healthysteps/)
- Treatment as usual (Active Comparator): DoD military treatment facility pediatric clinics follow American Academy of Pediatrics Bright Futures guidelines in providing well-baby care. The comparison arm of this study enrolled parents receiving treatment as usual under these guidelines at participating clinics assigned to this condition.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Other: HealthySteps (https://www.zerotothree.org/our-work/healthysteps/) — Within the DoD, most elements of the civilian HS model copyrighted by ZeroToThree.org were implemented. However, there were some modifications to accommodate the unique environment of the military community. The pilot utilized the pre-existing Military Family Life Counseling Program (MFLC) staff to serve as HS Specialists at participating clinics. MFLCs were hired and trained in the HS model through the HS Institute provided by ZeroToThree.org. Although the DoD pilot offered all 3 tiers of targeted care standard for the HS model, note that the DoD pilot did not offer a 24-hour parent support line at tier 1. Also, the DoD pilot required participating pilot clinics to utilize a modified version of the Tufts Survey of Well-Being of Young Children (SWYC; https://www.tuftsmedicine.org/medical-professionals-trainees/academic-departments/department-pediatrics/survey-well-being-young-children) to provide augmented screenings for infants at all tiers of pilot service provision.
  Arms: HealthySteps Pilot
Other: Treatment as Usual (TAU) — The comparison clinics included in this intervention were selected to represent pediatric care within military treatment facilities throughout the DHA medical system located at Army, Navy, Marine Corps, and Air Force facilities. There is variability in pediatric practice across military service branches. However, all clinics follow the American Academy of Pediatrics Bright Futures guidelines.
  Arms: Treatment as usual

SUMMARY:
BACKGROUND: The Defense Health Agency (DHA) and the Office of Military Community and Family Policy (MC&FP) requested assistance in evaluating the effectiveness of a military pilot implementation of a civilian program designed to assist families with infants called HealthySteps (HS; HealthySteps National Office, 2018). HS is a unique pediatric primary care-based program that helps families identify and manage parenting challenges. The program interweaves the medical support of the pediatrician's office with the resources and services of a HS Specialist trained to help parents understand their infants' needs (e.g., feeding, behavior, sleep) and their role as caregivers. HS Specialists provide enhanced educational support and facilitate targeted referrals to other relevant DoD and civilian support resources.

OBJECTIVE: The HS program has not been widely implemented or evaluated previously in a military context. However, a small 2-site pilot was initiated in 2017 by MC&FP to assess the feasibility of offering the HS program in military treatment facilities (MTF). The Defense Health Agency (DHA) further determined that this pilot program could be expanded to fulfill a 2019 National Defense Authorization Act (NDAA) requirement for the implementation and evaluation of a pilot program to reduce risk factors for child abuse and neglect within the U.S. military community.

APPROACH: This outcome evaluation study entailed a review of medical records for families enrolled in the HS pilot as well as the collection of prospective survey data. Survey data collected from primary caregivers enrolled in HS at seven implementation locations throughout the U.S. is being compared with survey data collected from caregivers of newborns seeking care at control locations offering pediatric treatment as usual.

VALUE: The HS program is expected to improve parental engagement in well-baby care, increase targeted screenings and referrals, improve parental efficacy and knowledge, as well as facilitate integration and utilization of existing family services available across disparate military support settings. It also is expected to increase military service satisfaction and perceived support among military parents. Summary reports of study results will be provided to MC&FP, DHA, and Congress.

RESEARCH COLLABORATORS: NHRC is a Department of the Navy Bureau of Medicine and Surgery research command located in San Diego, California. Abt Global is a leading civilian professional research corporation with extensive experience in military health research. Investigators from these two institutions are collaborating to conduct this outcome evaluation.

STUDY POPULATION: Participating pilot program clinics included 7 military pediatric clinic locations selected by DHA and serving personnel and their families from all U.S. military service branches. All families with children aged 0-4 months seeking well-baby care at participating MTF pilot pediatric clinics were eligible for HS program services and for study recruitment. Additionally, beneficiaries similarly seeking care for a newborn at 11 MTF pediatric clinics providing treatment as usual were eligible for the comparison condition. Medical records for this population were reviewed and prospective survey evaluation data were collected and merged together for ongoing analysis and reporting.

DETAILED DESCRIPTION:
The Defense Health Agency (DHA) and the Office of Military Community and Family Policy (MC&FP) requested assistance in evaluating the effectiveness of a military pilot implementation of the civilian, evidence-based program HealthySteps (HS; HealthySteps National Office, 2018). HS is a unique pediatric primary care-based program that helps families identify and manage parenting challenges through education and non-clinical counseling during pediatric visits. The program interweaves the medical support of the pediatrician's office with the resources and services of HS Specialists trained to help parents understand their infants' needs (e.g., feeding, behavior, sleep) and their role as caregivers. The Specialists provide enhanced educational support based on improved infant screening and facilitate targeted referrals to other DoD new parent support resources.

Under an approved NHRC Institutional Review Board protocol (NHRC.2019.0021), the study team conducted a 2-year prospective data collection recruiting caregivers eligible for the HS program at pilot implementation sites, as well as caregivers with newborns/infants enrolled for well-baby care under treatment as usual at comparison sites.

Within 30 days of HS pilot program launch, at participating pilot sites an initial announcement about the availability of services was emailed by DHA to all eligible families. Subsequently, MC&FP Military Family Life Counselors (MFLCs) serving at pilot sites as HS Specialists were provided with up-to-date lists of contact information for caregivers with initial well-baby visits at their clinic. Both families with newborns scheduling a first well-check and beneficiaries with infants up to 4 months of age transferring care from another clinic location were included in the contact lists. NHRC researchers also received copies of these lists. Contact information provided in these lists was used by Specialists to invite beneficiaries to receive pilot services and by the NHRC research team to recruit study participants. NHRC further requested similar contact lists for comparison sites to facilitate the use of comparable participant recruitment procedures at all participating locations.

DHA selected the original 7 sites that would participate actively in the HS pilot and 5 more to serve as comparison sites based on federal requirements outlined in NDAA FY19, section 578. At all of the original sites, NHRC conducted in-person data collection onsite. However, in order to ensure an adequate sample size and timely completion of baseline recruitment, NHRC further requested to receive weekly DHA contact lists for families receiving pediatric well-baby care as usual for infants aged 0-4 months at 6 additional Defense Health Agency MTFs. These additional locations were only engaged for remote (i.e., mail, email, phone) recruitment into the comparison condition.

The MTF pediatric clinics participating in the HS pilot program had some variability in the procedures HS Specialists were to follow in inviting families to take part in services and for enrolling them into the HS program. However, they were asked to enroll families--to the extent possible--at the time of the second well-baby check (2-weeks old). MC&FP provided all oversight for the implementation and staffing of the HS pilot services. However, the NHRC research team conducted a series of qualitative interviews with the pediatricians serving as primary points of contact for the pilot at each site in order to evaluate fidelity of program implementation.

The NHRC research team utilized flexible recruitment and data collection strategies in order to accommodate the requirements of each location. Across sites, NHRC recruited primary caregivers of newborns aged 0-4 months to maximize the dosage of HS services during the pilot evaluation (i.e., infants receive the most well-baby appointments over the course of the first year of life). Wherever possible NHRC also recruited families prior to their first engagement with the HS Specialists by enrolling them at the first clinic visit (2-3 days after birth). When engagement prior to the first HS visit was not possible, families were still recruited if they could be engaged prior to the second HS visit (2-month well-baby visit).

Because of the timing of the initiation of the outcome evaluation, a COVID-19 safety plan for NHRC data collectors was approved through the NHRC command. Researchers followed the command approved COVID-19 plan throughout the course of the study, as well as following any additional accommodations required by specific clinic sites. NHRC data collectors engaged families as soon as possible into the study, by attending newborn well-baby clinic visits held 2-3 days after birth. However, data collectors also were present to invite participants at other clinic appointments up to, but not including the 2-month visit. For families that the team could not contact at their 2-3 clinic visit, NHRC sent initial introductory invitation(s) via paper letter, phone message, and/or email with instructions for families to request a referral to the study through their pediatrician, clinic staff, or HS Specialist, by filling in their name and preferred mode of contact on a tear-off referral sheet and turning it in to one of these service providers. Furthermore, a poster and/or TV slides announcing the study were displayed in waiting areas at clinics where this was permitted. The study flyer was distributed to eligible families in clinic waiting rooms by clinic staff at time of intake. Families could request additional study information at any time by completing the flyer tear-off sheet and submitting it to a clinic staff member or giving it to an NHRC data collector. The flyer further included a QR code for the study website (www.dod-wellbabystudy.org) that listed procedures to submit requests for more study information as well; these web requests were received by the team via a study email address (usn.NHRC-HealthySteps@health.mil). Data collectors would then follow-up individually with these families using their preferred mode of contact to set up a phone or virtual meeting to explain more about the study.

Four types of data were collected for this study: 1) As part of study enrollment, contact information and demographics were collected on paper or pdf fillable forms 2) at three timepoints self-report survey data--excluding all identifiers except a random study ID number--were collected electronically on tablets, phones, or computers and transmitted over the internet to Abt Global for processing, 3) Specialists submitted HS program implementation records weekly to NHRC, and 4) archival administrative and medical data were extracted by NHRC and merged with self-report survey data for analysis. Survey data were collected at 1) baseline (defined as enrollment in the study), 2) six-months after baseline and 3) twelve-months after baseline. The archival data extracted from DHA patient health records and from Defense Manpower Data Center personnel records included identifiers, demographics, health records, and military career history information. HS implementation documentation records included an excel case management tracking record for each Specialist and pdf checklist forms for every HS visit where services were provided to eligible beneficiaries.

Follow-up data collection was conducted through remote (i.e., mail, email, phone) invitations and survey completion reminders sent by NHRC researchers approximately 6-months and 12-months after initial study enrollment. Up to three email invitations (approximately 2 weeks apart) and three postal mail invitations (approximately 2 weeks apart) were sent for each follow-up survey. If a participant enrolled in the study and began either a baseline or follow-up survey, but did not finish the survey immediately, the study team would send them survey completion reminders. Up to three emails (approximately 2 weeks apart) and three paper mailings (approximately 2 weeks apart) were sent until the time the participant completed their respective survey. In cases where the study team also had a participant's phone number, NHRC researchers would make up to 5 phone call attempts and leave up to 2 text messages and/or 2 voicemails (audio or text) reminding participants to complete their surveys. Participants receive a $20 downloadable gift code as an incentive after completing each of the three surveys.

Reports and briefings of study results are being shared with MC&FP, DHA, and with the U.S. Congress. Study results will provide these stakeholders with information regarding the impact of HS on multiple outcomes of interest. Implications for possible modification of the pilot or broader program implementation, based on evaluation results, also will be provided. Furthermore, the results will be disseminated to the community of military family researchers and service providers through presentation(s) and through publication(s) in academic venues.

Active study recruitment concluded June 30, 2023; and the baseline survey portal closed July 31,2023. The Study finalized follow-up data collection January 31, 2024. After January 31st when the survey portals closed, an explanatory message was posted on the study website in response to any attempts from prior participants or from the public to access the survey. The message noted that the study had concluded enrolling participants, and the study link was no longer available. It also instructed past participants to contact the study team (usn.NHRC-HealthySteps@health.mil) if they had any further questions.

ELIGIBILITY:
Inclusion Criteria:

* TRICARE eligible
* English-speaking
* Parent of an infant aged 0-4 months
* Seeking well-baby care at a participating military treatment facility pediatric clinic
* Expecting to be the caregiver most often attending well-baby appointments

Exclusion Criteria:

* Expecting to leave service or transfer locations/clinics within less than 6 months of WBWF enrollment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1181 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Well-baby care engagement | First year of infant's life
  We examined appointment file data in medical records for participating families to document well-child care (WCC) adherence. This was operationalized as the extent to which beneficiary caregivers brought their infants into the clinic for recommended well-child visits (Current Procedural Terminology codes 99381 and 99391). On-time well child visits were flagged using a classification strategy modeled after Goyal (2020) and based on a slightly modified version of the Bright Futures recommended periodicity (Bright Futures, 2024). Note that in DoD Pediatrics the recommended 1-month well-child check is scheduled early at 2 weeks. Expected timeframes were as follows: Visit1: 0-7 days; Visit2: 8-41 days; Visit3: 42-90 days; Visit4: 91-150 days; Visit5: 151-210 days; and Visit6: 211-335 days.
Timely vaccinations | First year of infant's life
  Adherence to infant vaccination schedules was evaluated as a benchmark metric for pilot program implementation success. The receipt of ten different pediatric vaccine series was documented from health records for infants at participating clinics, including Hepatitis A, Hepatitis B, Rotavirus, Diphtheria/Tetanus/Pertussis, Haemophilius Influenzae Type b, Pneumococcal Conjugate Vaccine, Polio, Measles/Mumps/Rubella, Varicella, and COVID. Using a classification strategy modeled after Romano et. al. (2022), Initial vaccine doses were considered on-time if they occurred prior to or no later than 4 days after the recommended age; similarly, follow-up doses were timely if they occurred prior to or no later than 4 days after the recommended interval. recommended vaccinations received within expected timeframes.
Emergency room visits | First year of infant's life
  We created an emergency room visit indicator documenting trips to the emergency room for infants in either the HS condition or control group conditions. Data for this indicator were extracted from archival medical records regarding medical encounters at MTF treatment facilities.
Social determinants of health | First year of infant's life
  Social determinants of health were evaluated using a modified 10-item version of the family needs assessment on the Tufts Survey of Well-being of Young Children (SWYC; Tufts Medicine, 2024). This section of the SWYC covers issues such as food insecurity, and parental well-being (e.g., substance use, marital quality/conflict). For the DoD HS pilot, participating pilot clinics were asked to use an augmented version of the SWYC family needs screener including 3 additional items regarding financial insecurity (i.e., housing, bills, and transportation). This augmented set of items was included on the WBWF study surveys at each time point. Note that as used in clinic screening and as a study outcome, total scores were not computed; rather a positive response to any of the 10 items was indicative of need.
Military life stress | First year of infant's life
  Based on a measure adapted from the Millennium Cohort Family Study (Corry, 2017; 2021), the WBWF asked parents regarding the stresses of military life, and in particular included a single item assessing the overall recent stress level ("In general, how stressful do you feel military life has been for you and your family over the past 6 months?" response options: 1 = not at all stressful to 5 = extremely stressful).
Parental depression | Infant's first year of life
  The Patient Health Questionnaire (Spitzer, 1999) 2-item screen for depression was used to asses for parental symptoms of depression at each survey timepoint. Respondents indicate the frequency of two key symptoms; (1) little interest or pleasure in doing things and (2) feeling down, depressed or hopeless. Responses options are on a 4-point scale ranging from "not at all" to "nearly every day." Higher total scores (range = 2 to 8) indicate more frequent symptomology.
Parenting quality: Attunement | Infant's first year of life
  The Attunement subscale of the Baby Care Questionnaire (Winstanley & Gattis, 2013) was used to assess the quality of participants parenting in caring for their newborns. Specifically, this subscale operationalizes parental sensitivity to infant cues and attentional states in parenting interactions. Scores on the Attunement subscale range from 0 to 70, with higher scores more clinically favorable.
Parenting quality: Structure | Infant's first year of life
  The Structure subscale of the Baby Care Questionnaire (Winstanley & Gattis, 2013) was additionally used to assess quality of parenting. This subscale operationalizes use of regularity and routines in infant care. Scores on the Structure subscale range from 0 to 85, with higher scores more clinically favorable.
Parenting competence: Efficacy | Infant's first year of life
  The Efficacy subscale from the Parenting Sense of Competence measure (Johnston & Mash, 1989) was used to assess new parents experiences in caring for their newborns, and in particular, their sense of instrumental competence, problem-solving ability, and capability in their caregiving role. Scores on the Efficacy subscale range from 0 to 28, with higher scores more clinically favorable.
Parenting Competence: Satisfaction | Infant's first year of life
  The Satisfaction subscale from the Parenting Sense of Competence measure (Johnston & Mash, 1989) was used to assess new parents experiences in caring for their newborns, and in particular, their sense of affective frustration, anxiety, and motivation in their caregiving role. Scores on the Satisfaction subscale range from 0 to 28, with higher scores more clinically favorable.
Augmented referrals | Infant's first year of life
  Improving processes for targeted referrals is a primary objective of the HS program and we assessed the percentage of families at HS pilot versus comparison locations receiving referrals to specific support services, including important military-specific support programs (e.g., DoD New Parent Support Program).
Work-family conflict | First year of infant's life
  Participants responded to 5 true/false items from the Work-Family Conflict Scale (Netemeyer et al., 1996) modified to apply to military life (e.g., my deployment-related travel [30 days or more] interferes with our home and family life). This measure was originally adapted for use in the Millennium Cohort Family Study. Response options were on a 5-point Likert type scale from 1 = strongly disagree to 5 = strongly agree (Sum scores range from 5-25, with higher scores indicating more conflict).
Infant difficulty | First year of infant's life
  A modified assessment of parent perceptions regarding how difficult their infant was to care for was included from the National Survey of Children's Health (Data Resource Center of Child and Adolescent Health, 2024). Scores from this 3-item subscale range from 0 to 12, with higher scores more unfavorable.
Protective factors: Family functioning | Infant's first year of life
  Family strengths and resources potentially protective against child maltreatment were assessed with the Protective Factors Survey (Counts, 2010) including a module regarding family functioning. Scores on this subscale range from 0 to 12, with higher scores more clinically favorable.
Protective factors: Nurturing and attachment | Infant's first year of life
  Family strengths and resources potentially protective against child maltreatment were assessed with the Protective Factors Survey (Counts, 2010) including a module regarding nurturing and attachment. Scores on this subscale range from 0 to 16, with higher scores more clinically favorable.
Protective factors: Social support | Infant's first year of life
  Family strengths and resources potentially protective against child maltreatment were assessed with the Protective Factors Survey (Counts, 2010) including a module regarding social support resources. Scores on this subscale range from 0 to 16, with higher scores more clinically favorable.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie A. Stander, Ph.D., Principal Investigator — Naval Health Research Center
Locations (2):
- United States (2):
  - Naval Health Research Center, San Diego, California
  - Abt Global, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] HealthySteps National Office. (2018). HealthySteps Implementation Guide. Author.
- [Background] Winstanley A, Gattis M. The Baby Care Questionnaire: a measure of parenting principles and practices during infancy. Infant Behav Dev. 2013 Dec;36(4):762-75. doi: 10.1016/j.infbeh.2013.08.004. Epub 2013 Sep 18. PMID 24050932
- [Background] Johnston C and Mash EJ. A measure of satisfaction and efficacy. (1989). Journal of ClinicalPsychology. 18 (2),167-175.
- [Background] Counts JM, Buffington ES, Chang-Rios K, Rasmussen HN, Preacher KJ. The development and validation of the protective factors survey: a self-report measure of protective factors against child maltreatment. Child Abuse Negl. 2010 Oct;34(10):762-72. doi: 10.1016/j.chiabu.2010.03.003. Epub 2010 Sep 19. PMID 20851466
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Netemeyer, R. G., Boles, J. S., & McMurrian, R. (1996). Development and validation of Work-Family Conflict and Family-Work Conflict Scales. Journal of Applied Psychology, 81(4), 400-410.
- [Background] Corry NH, Williams CS, Radakrishnan S, McMaster HS, Sparks AC, Briggs-King E, Karon SS, Stander VA. Demographic Variation in Military Life Stress and Perceived Support Among Military Spouses. Mil Med. 2021 Jan 25;186(Suppl 1):214-221. doi: 10.1093/milmed/usaa386. PMID 33499525
- [Background] Tufts Medicine. (2024). The Survey of Well-being of Young Children. Retrieved September 19 from https://www.tuftsmedicine.org/medical-professionals-trainees/academic-departments/department-pediatrics/survey-well-being-young-children
- [Background] Romano CJ, Bukowinski AT, Hall C, Burrell M, Gumbs GR, Conlin AMS, Ramchandar N. Brief Report: Pediatric Vaccine Completion and Compliance Among Infants Born to Female Active Duty Service Members, 2006-2016. MSMR. 2022 Nov 1;29(11):18-22. No abstract available. PMID 36790926
- [Background] Goyal NK, Rohde JF, Short V, Patrick SW, Abatemarco D, Chung EK. Well-Child Care Adherence After Intrauterine Opioid Exposure. Pediatrics. 2020 Feb;145(2):e20191275. doi: 10.1542/peds.2019-1275. Epub 2020 Jan 2. PMID 31896548
- [Background] Bright Futures. (2024). Recommendations for preventive pediatric health care. In Amer Acad of Pediatrics: Author.